CLINICAL TRIAL: NCT06131086
Title: Effect of Scapular Stabilization Exercises Along With Pectoralis Minor Stretching on Throwing Velocity of Male Fast Ballers Having Scapular Dyskinesia
Brief Title: Effect of Scapular Stabilization Excercise With Pectoralis Minor Stretching in Ballers Having Scapular Dyskinesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0456
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Scapular Dyskinesis; Pectoralis Minor Syndrome
Keywords: velocity; strenght; scapular stabilization

STUDY DESIGN:
Intervention Model Description: Randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the reading is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stabilization exercises (Experimental): Scapular stabilization exercise
  Scapular Retraction Exercise:
  2. Scapular Wall Slide: Stand with your back against a wall and your feet shoulder-width apart.Raise your arms to shoulder height with your elbows bent at a 90-degree angle, so that your hands are pointing up
  * Slide your arms up the wall as high as you can, while keeping your shoulder blades pinched together and down
  * Hold the position for 5-10 seconds, then slowly lower your arms back down to the starting position
  * Repeat for 10-15 repetitions
  Interventions: Other: stabilization exercises
- stabilization exercises along with pectoralis minor stretching (Experimental): pectoralis minor stretch: Stand facing a wall or a doorway. Raise your right arm to shoulder height and place your right forearm against the wall or doorway, with your elbow bent at a 90-degree angle.
  Step forward with your right foot until you feel a stretch in your chest and shoulder.
  Slowly lean forward, keeping your arm against the wall or doorway, until you feel a deeper stretch in your chest and shoulder.
  Hold the stretch for 10-15 seconds, then release and repeat on the other side. Repeat the stretch 2-3 times on each side.
  Interventions: Other: stabilization exercises along with pectoralis minor stretching

INTERVENTIONS:
Other: stabilization exercises — this include stabilization exercise thrice a week for six weeks
  Arms: stabilization exercises
Other: stabilization exercises along with pectoralis minor stretching — this include stabilization exercise with pectoralis minor thrice a week for six weeks
  Arms: stabilization exercises along with pectoralis minor stretching

SUMMARY:
The study is randomized and single -blinded. Ethical approval is taken from ethical committee of Riphah International university Lahore. participant selected through non probability convenience sampling technique on 26 fast bowlers which further players were randomly divided into two groups, group A (Experimental group) and group B (Control group), having 13 players in each group. Scapular stabilization exercises along with pectoralis minor stretching were administered in group A whereas generalized shoulder exercises along with self-stretching of shoulder muscles were performed in group B.

DETAILED DESCRIPTION:
It will be randomized controlled trial (RCT) research design at AL Fatah sports complex and Saeed Ajmal cricket academy through non probability convenience sampling technique on 26 fast bowlers which further players were randomly divided into two groups, group A (Experimental group) and group B (Control group), having 13 players in each group. Scapular stabilization exercises along with pectoralis minor stretching were administered in group A whereas generalized shoulder exercises along with self-stretching of shoulder muscles were performed in group B. Assessment will be made by pocket radar, pectoralis minor index and Vernier caliper. There will be 3 sessions in a week for 6 weeks. The baseline scoring will be on 1st day, follow up will be taken at 6th week. Data will be analyzed during SPSS software version 26. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

Male fast ballers

* 21-30 years of age
* Duration of playing at least 1 to 2 years
* Dominant side effected

Exclusion Criteria:

* • Old fracture at effected arm

  * Any serious injury during treatment
  * Patient with cervical spondylosis and neurological abnormalities at effected arm

Ages: 21 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
velocity | pre and 6 weeks post interventional
  will be measured by pocket radar
pect minor length | pre and 6 weeks post interventional
  will be measured by pectoralis minor lenght

CONTACTS AND LOCATIONS:
Overall Officials: usman ali, DPT, Principal Investigator — Investigator
Locations (1):
- Al fatah sport complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnorenberg AJ, French ME, Riebe JM, Grindel SI, Slavens BA. Shoulder complex kinematics pre- and post- rotator cuff repair. J Electromyogr Kinesiol. 2022 Feb;62:102331. doi: 10.1016/j.jelekin.2019.07.001. Epub 2019 Jul 2. PMID 31324512
- [Background] Longo UG, Risi Ambrogioni L, Berton A, Candela V, Massaroni C, Carnevale A, Stelitano G, Schena E, Nazarian A, DeAngelis J, Denaro V. Scapular Dyskinesis: From Basic Science to Ultimate Treatment. Int J Environ Res Public Health. 2020 Apr 24;17(8):2974. doi: 10.3390/ijerph17082974. PMID 32344746
- [Background] Blache Y, Begon M, Michaud B, Desmoulins L, Allard P, Dal Maso F. Muscle function in glenohumeral joint stability during lifting task. PLoS One. 2017 Dec 15;12(12):e0189406. doi: 10.1371/journal.pone.0189406. eCollection 2017. PMID 29244838
- [Background] Kibler WB, Sciascia A. Evaluation and Management of Scapular Dyskinesis in Overhead Athletes. Curr Rev Musculoskelet Med. 2019 Dec;12(4):515-526. doi: 10.1007/s12178-019-09591-1. PMID 31760624
- [Background] Sterling M. Physiotherapy management of whiplash-associated disorders (WAD). J Physiother. 2014 Mar;60(1):5-12. doi: 10.1016/j.jphys.2013.12.004. Epub 2014 Apr 24. No abstract available. PMID 24856935
- [Background] Nunes MK, Fontenele Dos Santos G, Martins E Silva DC, Mota de Freitas AC, Henriques IF, Andrade PM, Machado Dde C, Teixeira S, Neves MO, Dias G, Silva-Junior F, Bastos VH. Acute effects of neural mobilization and infrared on the mechanics of the median nerve. J Phys Ther Sci. 2016 Jun;28(6):1720-3. doi: 10.1589/jpts.28.1720. Epub 2016 Jun 28. PMID 27390402